CLINICAL TRIAL: NCT04432233
Title: Intravenous Administration of Metronidazole, Levofloxacin and Esomeprazole Triple Therapy in the Treatment of Helicobacter Pylori Infection and Related Complications Caused by Active Peptic Ulcer Disease
Brief Title: Intravenous Triple Therapy in the Treatment of Helicobacter Pylori Infection and Related Complications Caused by Active Peptic Ulcer Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rjkls2020031
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Helicobacter Pylori Infection; Intravenous Drug Usage
Keywords: Helicobacter Pylori Infection; Intravenous Drug Usage
MeSH Terms: interventions — Esomeprazole; Metronidazole; Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intravenous therapy (Experimental): Subjected enrolled will receive (a) a 10-day intravenous triple therapy containing esomeprazole 40 mg thrice a day, metronidazole 500 mg twice a day and levofloxacin 500 mg once a day and (b) esomeprazole 20 mg twice a day taken orally for 8 weeks.
  Interventions: Drug: Esomeprazole; Drug: Metronidazole; Drug: Levofloxacin

INTERVENTIONS:
Drug: Esomeprazole — Proton pump inhibitor
Drug: Metronidazole — antibiotic for H. pylori eradication
Drug: Levofloxacin — antibiotic for H. pylori eradication

SUMMARY:
Helicobacter pylori infection causes active peptic ulcer disease and related complications like bleeding and pyloric obstruction. Usually, clinicians tended to treat Helicobacter pylori infection after active peptic ulcer disease and related complicaitons getting healed, which spent time and money. This study is designed to evaluate the efficacy and safety of intravenous administration of metronidazole, levofloxacin and esomeprazole triple therapy in the treatment of Helicobacter pylori infection combined with peptic ulcer disease related complications.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 75 years old
* Without previous Helicobacter pylori treatment
* Diagnosed with active peptic ulcer disease and related complications like bleeding and pyloric obstruction by endoscopy examination
* Ability and willingness to participate in the study and to sign and give informed consent
* Positive for Helicobacter pylori IgM antibody

Exclusion Criteria:

* With previous gastric surgery
* Major systemic diseases
* Pregnancy or lactation
* Allergy to any of the study drugs
* Decline to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Six weeks after completion of therapy
  Six weeks after completion of therapy, H. pylori eradication was assessed by ¹³C-urea breath test. Eradication was defined as negative result from urea breath test (<4‰) (4‰ as the cutoff value).

SECONDARY OUTCOMES:
Rate of adverse effects | Within 7 days after completion of therapy
Rate of stop bleeding | Within 7 days after completion of therapy
Rate of pyloric obstruction remission | Within 7 days after completion of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Hong Lu, PHD,MD, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No